CLINICAL TRIAL: NCT02820831
Title: Anesthesia Geriatric Evaluation and the Prediction of Quality of Life in Elderly Peripheral Vascular Surgery Patients
Brief Title: Anesthesia Geriatric Evaluation and Quality of Life After Peripheral Vascular Surgery
Acronym: AGE-VASC
Status: Terminated | Type: Observational
Why Stopped: Slow inclusion
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, dr. P.G. Noordzij, St. Antonius Hospital
Other Study IDs: NL 55038.100.15
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life
Keywords: Frail Elderly; Peripheral Vascular Surgery; Risk Assessment; Functional status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are taken directly after induction of anesthaesia. Plasma is stored in frozen aliquots at - 80 degrees Celcius.

SUMMARY:
A prospective observational cohort study to assess the predictive value of preoperative frailty on postoperative quality of life in peripheral vascular surgery patients.

DETAILED DESCRIPTION:
Introduction:

The percentage of elderly in the general population is increasing rapidly. Currently, the Dutch population comprises for one fifth of persons aged 65 years or older and recent estimates show this will increase to roughly a quarter in the next 20 years. Since th incidence of peripheral arterial disease increases with age, this rise in elderly will also reflect on the population of patients being referred for vascular surgery. Elderly patients are at higher risk for postoperative complications, mortality or functional decline than younger patients. In frail elderly this effect might be more pronounced. Frailty is an umbrella term that encompasses patient related factors such as weight loss, muscle wasting, inactivity, comorbidities and polypharmacy. Current scoring systems that are used to predict postoperative mortality and complications following vascular surgery perform poorly in the elderly population and do not take into account frailty. Moreover they are designed to predict mortality and complications and are not validated to predict patient reported outcome measures such as quality of life or functional status. The aim of the AGE VASC study is assess the value of frailty factors in predicting an improvement in quality of life one year after peripheral vascular surgery.

Methods:

The AGE VASC study is a prospective observational cohort study. All patients aged 70 years or older, scheduled for peripheral vascular surgery of the lower limb, mentally competent and have signed informed consent are eligible for the study. Before surgery patients will be screened for frailty using different questionnaires and physical tests. The battery of tests exists of Short Form 36 (SF36), Walking Impairment Questionnaire (WIQ), Multi Nutritional Assessment (MNA), Montreal Cognitive Assessment (MoCA), Nagi's scale for disability, Geriatric Depression Scale -8 (GDS8), three physical tests: five meter walking speed, timed get up and go test and hand grip strength. And a non-invasive measurement of Advanced Glycation Endproducts (AGEs). A blood sample will be taken to determine vitamin status, immune status and iron deficiency. After surgery, electronic patients charts will be studied to score postoperative complications or mortality. Three and twelve months after surgery patients will receive SF-36, WIQ, and World Health Organization Disability Assessment Schedule (WHODAS) 2.0 questionnaires to determine quality of life and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or older
* Mentally competent
* Planned peripheral vascular surgery of the lower limb (femoral artery desobstruction, bypass surgery, amputation), possibly combined with endovascular procedure
* Signed informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients planned for elective vascular surgery of the lower limb or amputation including surgical procedured combined with endovascular.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 12 months after surgery
  Assessed by Medical Outcomes Study Short Form-36 (SF-36)

SECONDARY OUTCOMES:
Quality of Life | 3 months after surgery
  Assessed by Medical Outcomes Study Short Form-36 (SF-36)
Walking Impairment | 3 and 12 months after surgery
  Assessed by Walking Impairment Questionnaire
Psychosocial or physical functioning | 3 and 12 months after surgery
  Assessed by World Health Organisation Disability Assessment Schedule 2.0 (WHODAS 2.0)
Incidence of postoperative complications and mortality | 30 days after surgery
  Postoperative complications scored are mortality, rebleed, infection, hematoma, respiratory insufficiency, cerebrovascular accident, renal failure.
Length of in-hospital stay | Post-surgical. The expected length of stay is 5-7 days
  Length of stay will be measured from date of surgery to date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Noordzij, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius hospital, Nieuwegein, Utrecht, Netherlands